CLINICAL TRIAL: NCT00990002
Title: INVESTIGATION OF CHANGES IN LEUKOCYTE POPULATIONS AMONG CHILDREN RECEIVING A FOLLOW-ON COW'S MILK-BASED FORMULA CONTAINING DIFFERENT BIOACTIVE INGREDIENTS.
Brief Title: Investigation of A Children's Beverage Containing Different Probiotics
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Collaborators: Father Flanagan's Boys' Home (Other)
Responsible Party: Bryan Liu, Mead Johnson Nutrition
Other Study IDs: 6002
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: A children's milk-based beverage
- experimental probiotic 1: children's milk-based beverage containing a bioactive ingredient
- experimental probiotic 2: children's milk-based beverage containing a different bioactive ingredient

SUMMARY:
Investigating different bioactive ingredients in children's beverages and the effect on blood serum markers.

ELIGIBILITY:
Inclusion Criteria:

* Children 2-4 years of age, weight and length for age within the 10th to 90th percentiles as plotted on the NCHS growth chart
* Consuming cow's milk for at least one month

Exclusion Criteria:

* Serious concurrent illness or acute infection
* Using systemic antibiotics or steroids
* Recent probiotic use
* Feeding difficulties or intolerance to cow's milk
* Conditions effecting normal growth and development
* Immunodeficiencies

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children 2-4 years of age
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Boys Town National Research Hospital, Boys Town, Nebraska, United States